CLINICAL TRIAL: NCT05336344
Title: Supporting Family Caregivers of Persons With Dementia
Acronym: ENCODE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, George Demiris, PhD, PIK University Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 849217
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Caregiver Stress Syndrome; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Clinical Coding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENCODE Group (Experimental): The intervention consists of three weekly video-conferencing sessions scheduled at the caregiver's convenience. Each session is scheduled to last approximately 40 minutes. The ENCODE intervention is manualized and has related curriculum designed specifically for caregivers of patients with ADRD. The agenda for the first session (week 1) includes an assessment of caregivers' pain management challenges and concerns. Once the barriers or challenges are identified, the interventionist works specific problem solving therapy steps covered over the three sessions.
  Interventions: Behavioral: ENCODE
- Attention Control Group (No Intervention): Caregivers in the attention control group will receive standard hospice services and complete the same measures and receive the same number of contacts as participants in the intervention group. Three video-conferencing calls will be scheduled based on the caregiver's availability following, if possible, a timeline between days 5 and 30 of the hospice admission. During these calls, the interventionist will allow caregivers in the attention control group to discuss their feelings, thoughts, and relationships. This "friendly call" intervention controls for the nonspecific aspects of treatment, i.e., the passage of time, amount of contact with a researcher, and the general support of an empathic, concerned and skilled professional and is based on the principles of nondirective supportive therapy.

INTERVENTIONS:
Behavioral: ENCODE — a cognitive behavioral intervention for family caregivers to improve pain management skills and overall coping
  Arms: ENCODE Group

SUMMARY:
Based on preliminary work, whereby investigators examined pain management challenges and needs of caregivers of hospice patients with dementia, this team designed a cognitive behavioral intervention informed by the relational model of stress, entitled ENCODE (Empowering Caregivers of Patients with Dementia) to assist caregivers in effectively identifying and communicating their pain management challenges and needs. The investigators propose a 5-year randomized clinical trial in which caregivers of patients with Alzheimer's Disease and Related Dementias (ADRD) will be randomly assigned to a group receiving standard hospice care with the addition of "friendly video-calls" providing social support (attention control group) or a group receiving standard hospice care with the addition of the ENCODE intervention (intervention group).

DETAILED DESCRIPTION:
According to a report by the National Hospice and Palliative Care Organization published in 2020, over 180,000 Americans with a primary diagnosis of Alzheimer's disease or related dementias (ADRD) received hospice care in the United States in 2018. Although many of these patients and their families receive high quality care, numerous health care professionals have observed shortfalls in hospice care for patients with dementia, especially in the area of pain management. Past studies have shown a mixed impact of hospice enrollment on pain management for patients with ADRD. Shega et al found that roughly half of caregivers reported moderate or severe pain for patients with dementia, irrespective of hospice enrollment.

Core to the hospice philosophy is the goal to reduce or even eliminate suffering in patients and to support and address the needs of both patients and their families. Family caregivers, namely family and friends who provide informal, unpaid care to hospice patients, are essential to the delivery of hospice services; however, most lack formal healthcare training. A typical family caregiver of a hospice patient with ADRD will spend at least 46 hours per week assisting with activities of daily living, including personal hygiene, medication management, household chores, and transportation. Informal caregivers are 'on call' 24 hours a day and at high risk for chronic stress, deteriorating physical health, financial difficulties, and premature death. Informal caregivers suffer from high rates of depression and anxiety, and in the few studies that have focused on their experiences, pain management has been the most commonly expressed concern. Several studies have highlighted that challenges in communication about pain among patients, caregivers and clinicians is a major struggle for family caregivers; understanding the origin of this difficulty could lead to improvements in caregiver training and support. Many caregivers report feeling stressed about pain management and describe clinicians' strategies for pain management in ADRD care as "mysterious" or "suspicious".

In the general population of older adults with ADRD, attempts to precisely estimate the prevalence of pain and quality of pain management have met with varied success. One study of long-term dementia care units found that 18% to 30% of patients self reported pain, but prevalence of pain jumped to 50% when behavioral observation scales were used. Self-report of pain is limited in patients with advanced dementia, and the etiology of pain difficult to determine. In addition, patients may resist pain treatments due to their inability to understand the purpose of analgesia and may receive decreased benefit from analgesia due to the disruption of the placebo effect. Pharmaceutical pain treatments may also exacerbate symptoms of dementia such as agitation and confusion.

Based on preliminary work, whereby the investigators examined pain management challenges and needs of caregivers of hospice patients with dementia, the team designed a cognitive behavioral intervention informed by the relational model of stress, entitled ENCODE (Empowering Caregivers of Patients with Dementia) to assist caregivers in effectively identifying and communicating their pain management challenges and needs. The investigators recently completed a single group pilot study of the ENCODE intervention that demonstrated feasibility, acceptability and preliminary efficacy on improving caregiver quality of life and reducing anxiety. This study proposes a 5-year randomized clinical trial in which caregivers of patients with ADRD will be randomly assigned to a group receiving standard hospice care with the addition of "friendly video-calls" providing social support (attention control group) or a group receiving standard hospice care with the addition of the ENCODE intervention (intervention group). The specific aims are:

Aim 1: To assess the impact of the ENCODE intervention on caregiver quality of life (primary outcome) and caregiver anxiety, depression, health and caregiver's perception of patient pain (secondary outcomes).

Hypothesis 1a: Caregivers in the intervention group will report higher levels of (covariate-adjusted) post intervention quality of life compared to caregivers in the attention control group.

Hypothesis 1b: Caregivers in the intervention group will report higher levels of (covariate-adjusted) post intervention health, and lower levels of (covariate-adjusted) anxiety and depression and patient pain compared to caregivers in the attention control group.

Aim 2: To assess caregivers' perceptions of and satisfaction with the ENCODE intervention.

Aim 3: To facilitate the translation of the intervention into practice, and more specifically:

Aim 3a: conduct an analysis comparing costs associated with the control and the intervention groups.

Aim 3b: identify barriers and facilitators to adoption of a behavioral intervention aiming to facilitate pain management in hospice

ELIGIBILITY:
Inclusion Criteria:

* enrolled as a family/informal caregiver of a hospice patient with primary or secondary diagnosis of Alzheimer's disease or other related dementia
* responding with "yes" to the question about having any concerns about effectively managing their care recipient's pain
* 18 years or older
* no or only mild cognitive impairment
* speak and read English, with at least a 6th-grade education

Exclusion Criteria:

* Significant hearing loss that does not allow the participant to conduct telephone conversations as assessed by the research staff (by questioning and observing the caregiver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Caregiver Quality of Life-Index (CQLI-R) scores | assessments at week 1, week 3 and 40 day follow-up
  The CQLI-R, a four-item measure of caregivers' quality of life (QOL), includes four dimensions: emotional, social, financial, and physical. Total score ranges from 0 to 40 (higher score indicates higher quality of life).

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder (GAD-7) for caregivers | assessments at week 1, week 3 and 40 day follow-up
  The GAD-7 is a brief, valid tool for screening for GAD and assessing its severity in clinical practice and research. The total score is calculated by assigning scores of 0-3 for each of the seven items. Scores of 5, 10, and 15 are taken as the cut off points for mild, moderate, and severe anxiety, respectively. The GAD-7 score ranges from 0 to 21, higher score indicates higher level of anxiety.
Change in the Depression Scale of the Patient Health Questionnaire (PHQ-9) | assessments at week 1, week 3 and 40 day follow-up
  The PHQ-9 is a nine-item tool for assessing and monitoring levels of depression. It assesses symptoms and functional impairment due to depression and derives a severity score. A higher score indicates higher level of depression. A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression
Change in the Pain Assessment in Advanced Dementia (PAINAD) Scale score | assessments at week 1, week2, week 3 and 40 day follow-up
  The PAINAD is a simple, valid, and reliable instrument for measurement of pain in noncommunicative patients with dementia. Unlike other scales developed for non-communicative patients that require extensive training and can only be administered by clinicians, PAINAD can be completed by caregivers themselves; it includes five items (breathing independent of vocalization, negative vocalization, facial expression, body language and consolability) generating a total score ranging from 0 to 10. A higher score indicates higher level of patient pain as assessed by the caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate de-identified data may be shared with other researchers upon a Data Use Agreement.